CLINICAL TRIAL: NCT03820960
Title: Risk Factors for Thrombosis in Immune Thrombocytopenia
Acronym: RiFT-ITP
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0148
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Immune Thrombocytopenia
Keywords: Thrombosis
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune thrombocytopenia (ITP) is a rare autoimmune disease (annual incidence: 3-4/105 inhabitants) leading to an increased risk of spontaneous bleeding. ITP is said "primary" when not associated to other systemic disease (lymphoma, systemic autoimmune disease, chronic infectious disease…). First-line treatment is based on corticosteroids. Intravenous immunoglobulin (IVIg) is added in case of serious bleeding. In about 70% of adult cases, ITP becomes persistent or chronic (lasting >3 months and >12 months, respectively). Second-line treatments are then indicated. Among them, thrombopoietin-receptor agonists (TPO-RAs), romiplostim and eltrombopag are increasingly used. Splenectomy is used as ultimate treatment.

Paradoxically, the risk of thrombosis is higher in ITP patients in comparison with the general population, due to the release of young hyperactive platelets from bone marrow. The incidence of thrombosis in ITP patients has been estimated between 0.5 and 3/100 patients-years. However, risk factors for thrombosis in ITP are not known, except splenectomy that is used in very few patients now. The role of other ITP treatments in thrombosis occurrence has been evoked, particularly for corticosteroids and IVIg. TPO-RAs have been associated with a risk of thrombosis in clinical trials and pharmacovigilance studies, even in case of low or normal platelet count. However, this risk has not been measured in the real-life practice, adjusted for other risk factors for thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Incident primary ITP adults

Exclusion Criteria:

* Secondary as well as prevalent ITP patients on July, 30th 2009 are excluded by the algorithm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational population-based study in France in the French Adult Immune THrombocytopenia (FAITH) cohort from July 2009 until June 2015. The FAITH study identifies since July 2009 all incident primary ITP adults in France within the national health insurance database (Système National d'Informations Inter-Régimes de l'Assurance Maladie, SNIIRAM, >66 million inhabitants).
Sampling Method: Non-Probability Sample
Enrollment: 10039 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Risk for thrombosis in adult primary ITP patients treated with ITP treatment | from July 2009 until June 2015
  Number of first hospitalization for arterial and veinous thrombosis in patients treated with ITP treatment

SECONDARY OUTCOMES:
Risk thrombosis in adult primary ITP patients treated with TPO-RAs. | from July 2009 until June 2015
  Number of first hospitalization for arterial and veinous thrombosis in patients treated with ITP patients treated with TPO-RAs.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Moulis, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

REFERENCES:
- [Result] Lafaurie M, Maquet J, Baricault B, Ekstrand C, Christiansen CF, Linder M, Bahmanyar S, Norgaard M, Sailler L, Lapeyre-Mestre M, Sommet A, Moulis G. Risk factors of hospitalisation for thrombosis in adults with primary immune thrombocytopenia, including disease-specific treatments: a French nationwide cohort study. Br J Haematol. 2021 Nov;195(3):456-465. doi: 10.1111/bjh.17709. Epub 2021 Aug 12. PMID 34386974